CLINICAL TRIAL: NCT06756997
Title: The Effect of Different Sensory Conditions on Sensory Interaction in Balance
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Assistant Professor, Dr., Bezmialem Vakif University
Other Study IDs: E-54022451-050.04-173777
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: Balance Assessment; Sensory Science
Keywords: balance assessment; sensory condition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group: Healthy Young Adults

SUMMARY:
The ability of humans to maintain spatial orientation and balance control relies on accurate and complete sensory information. This study aims to investigate the effects of different sensory conditions on the sway index (balance). Adults with normal hearing, vision, and balance abilities will perform the Modified Clinical Test of Sensory Interaction on Balance (mCTSIB), a test from the Biodex Balance System, under varying sensory conditions. The first sensory condition involves situations where the cursor indicating the individual's center of gravity on the device is either visible or hidden. The second condition examines whether the eyes-closed state during the test is achieved through voluntary eye closure or by external equipment (e.g., goggles or eye patches). The values obtained will allow comparisons of the effects of different sensory conditions on the sway index. The study will be conducted between January 2025 and March 2025 at the Bezmialem Vakıf University Cardiac Physiotherapy and Rehabilitation Education and Research Laboratory with healthy young adults. Participants will be selected voluntarily, and the assessments will be conducted in compliance with the guidelines of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 45.
* Providing informed consent to participate in the study after receiving detailed information about the research.

Exclusion Criteria:

* Having visual or hearing impairments.
* Presence of musculoskeletal, neurological, or orthopaedic conditions (e.g., lower extremity alignment disorders, excessive anteversion, severe pes planus) that could affect the study results.
* Having mental or physical problems severe enough to impair communication.
* Participation in any rehabilitation program within the past six months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the study will consist of 23 volunteer healthy young adult subjects aged 18-45 years. All subjects will be evaluated and tested at Bezmialem Vakif University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) | "From January 2025 to February 2025
  The assessment of postural control will be conducted using the Biodex Balance System® (BBS) (Biodex Medical Systems, Shirley, New York, USA). The BBS consists of a balance platform, handrails, a display, and a printer, it is a computer-assisted device with established validity and reliability, used to evaluate postural stability, limits of stability, and fall risk.
  The device features a movable platform capable of providing surface tilts up to 20˚ and a 360˚ range of motion, allowing individuals to move forward, backwards, left, and right. By altering the platform's tilt and range of motion, the difficulty level of the test can be adjusted. Mobility levels range from 1 (minimum) to 12 (maximum).
  This test evaluates how different sensory systems contribute to balance and assesses an individual's ability to compensate when one or more sensory inputs are compromised. The tests will be performed in the following sequence, and the sway index will be calculated for each test conducted.
Assessment Form | "From January 2025 to February 2025
  The "Assessment Form" will be used to record the demographic and medical history information of the healthy adult participants included in the study. The assessment form includes demographic details such as name, surname, gender, age, occupation, dominant side, and educational level, as well as medical and family history and the BBS assessment form.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided